CLINICAL TRIAL: NCT00970892
Title: Evaluation of VKORC1 and Cytochrome P450 CYP2C9 Gene Polymorphisms and Management of Warfarin Dose Using Pharmacogenetic Data
Brief Title: VKORC1 and CYP2C9 Gene Polymorphisms and Warfarin Management
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ankara University (Other)
Responsible Party: NEJAT AKAR, Prof., Ankara University
Other Study IDs: B.30.2.ANK.0.20.05.04
Record Dates: First submitted 2009-09-02; First posted 2009-09-03 (Estimated); Last update posted 2009-09-03 (Estimated); Status verified 2009-09

CONDITIONS: Atrial Fibrillation; Cardiac Thrombus; Deep Vein Thrombosis; Pulmonary Embolism; Heart Valve Replacement (Mechanical or Biological With AF); Cardiomyopathy (Ischemic or Dilated); Peripheral Vascular Disease
Keywords: Anticoagulation; warfarin; VKORC1; CYP2C9; thromboembolism; pharmacogenetics
MeSH Terms: conditions — Atrial Fibrillation; Venous Thrombosis; Pulmonary Embolism; Cardiomyopathies; Ischemia; Dilatation, Pathologic; Peripheral Vascular Diseases; Vitamin K-Dependent Clotting Factors, Combined Deficiency Of, Type 2; Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Warfarin dose titration — Dosage

SUMMARY:
The investigators aimed to use pharmacogenetic information in clinical practise which may lead to rapid, efficient, and safe warfarin dosing in this observational prospective study. In this context, the investigators plan to develop an algorithm for estimating the appropriate warfarin dose that is based on both clinical and genetic data from the Turkish study population. This study is unique not only investigating clinical factors, demographic variables, CYP2C9, and VKORC1 gene variations which contribute to the variability among patients in dose requirements for warfarin but also including thrombogenic single nucleotide polymorphisms (SNP) in the same patient population. Thus, warfarin would be a good example by being the first cardiovascular drug for pharmacogenetic guided "personalized medicine" applications.

DETAILED DESCRIPTION:
Long-term anticoagulation therapy with warfarin is recommended for patients with atrial fibrillation/flutter (AF), left atrial thrombus, deep vein thrombosis (DVT), pulmonary thromboembolism (PE), mechanical heart valve replacement, cardiomyopathy, and ischemic stroke. Warfarin, a coumarin derivative, produces an anticoagulant effect by interfering with the vitamin K 2,3 epoxide reductase (VKOR) enzyme and γ-carboxylation of vitamin K-dependent clotting factors such as II, VII, IX, and X. However, management of warfarin therapy is complicated with interindividual differences in drug response, delayed onset of action, difficulty with reversal and a narrow therapeutic window leading to increased risk of life-threatening hemorrhagic adverse events or thromboembolism. Furthermore, in order to determine safe and effective loading dose during the early phase of therapy and maintenance doses require frequent laboratory monitoring and adjustments to compensate for changes in patients' age, body size, vitamin K intake through diet, disease state, comorbidities, concomitant use of other medications, and patient-specific genetic factors.

Poor anticoagulant control may cause fatal complications such as thromboembolism with undertreatment or bleeding with excessive anticoagulation. Indeed, the risk of major bleeding in patients on warfarin is between 1% and 5% per year. Identifying the optimal therapeutic range and managing the dose of therapy to achieve the maximal time in therapeutic range are two of the most important determinants of therapeutic effectiveness and of reducing hemorrhagic risk. Currently, there have been substantial efforts to improve the safety of warfarin anticoagulation therapy. Recent warfarin pharmacogenetic studies have largely focused on two candidate genes: CYP2C9, responsible for warfarin metabolism, and VKORC1, which encodes vitamin K epoxide reductase, the site of warfarin action. Current evidence is clear that polymorphisms in either CYP2C9 or VKORC1 affect warfarin sensitivity.

We aimed to use pharmacogenetic information in clinical practise which may lead to rapid, efficient, and safe warfarin dosing in this observational prospective study. In this context, we plan to develop an algorithm for estimating the appropriate warfarin dose that is based on both clinical and genetic data from the Turkish study population. This study is unique not only investigating clinical factors, demographic variables, CYP2C9, and VKORC1 gene variations which contribute to the variability among patients in dose requirements for warfarin but also including thrombogenic single nucleotide polymorphisms (SNP) in the same patient population. Thus, warfarin would be a good example by being the first cardiovascular drug for pharmacogenetic guided "personalized medicine" applications.

ELIGIBILITY:
Inclusion Criteria:

Patients who require warfarin for at least 6 months with the indications listed below:

* Permanent Atrial Fibrillation/Flutter
* Left atrial or ventricular thrombus
* Deep Vein Thrombosis
* Pulmonary Embolism
* Heart Valve Replacement (Mechanical or Biological With AF)
* Cardiomyopathy (Ischemic or Dilated)
* Peripheral Vascular Disease

Exclusion Criteria:

* History of GI bleeding or peptic ulcer disease
* Significant liver disease, active hepatitis or chronic HBV/HCV infection
* Uncontrolled hypertension
* Chronic diarrhea or malabsorption syndrome
* Viral or bacterial infection prior to enrollment
* Active or previous infective endocarditis
* Hospital stay > 30 days as a result of septicemia, mediastinitis or pneumonia
* Cardiac cachexia
* Morbid obesity
* Expected pregnancy, pregnancy or lactation
* Psychiatric disease
* Malignancy with Life expectancy less than 1 year

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who require warfarin for at least 6 months under care of cardiovascular surgery, cardiology and pulmonary disease.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2009-07; Primary Completion 2012-07 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Warfarin related complications including bleeding and thromboembolism | 6 months

SECONDARY OUTCOMES:
Maximal time in international normalized ratio (INR) therapeutic range and deviation from target INR levels | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Nejat Akar, Prof, Principal Investigator — Ankara University
Locations (1):
- Ankara University Medical Faculty, Department of Cardiovascular Surgery and Pulmonary Disease, Ankara, Turkey (Türkiye)